CLINICAL TRIAL: NCT03202173
Title: The Diagnosis of the Squamous Cell Carcinoma in Head and Neck by Using the Probe-based Confocal Laser Endomicroscopy
Brief Title: The Diagnosis of NPC Using the Probe-based Confocal Laser Endomicroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Huawei Li, Ph.D, MD, Director of Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Eye & ENT Hospital of Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: pCLE in the diagnosis of NPC
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Nasopharyngeal Carcinoma; Squamous Cell Carcinoma of the Head and Neck
Keywords: Probe-based confocal laser endomicroscopy; Optical biopsy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal mucosa (Active Comparator): Flat and relatively uniform polygonal epithelial cells with alternating dark and light bands were noted in pCLE images of normal mucosa after intravenous injecting 10% fluorescein.
  Interventions: Diagnostic Test: 10% fluorescein
- lymphoid hyperplasia (Experimental): An unorganized tissue architecture, irregular cells (difference of cell shape, color and size), slightly intensified fluorescein leakage, and vessels not assessable were found in the lymphoid hyperplasia of nasopharyngeal mucosa after intravenous injecting 10% fluorescein..
  Interventions: Diagnostic Test: 10% fluorescein
- nasopharyngeal carcinoma (Experimental): pCLE images of nasopharyngeal carcinoma, which was associated with crowded unorganized tissue architecture (a dark-gray background without identification of mucosal structures), irregular cells like cell clusters, amplified fluorescein leakage, and irregular vessels changes after intravenous injecting 10% fluorescein.
  Interventions: Diagnostic Test: 10% fluorescein

INTERVENTIONS:
Diagnostic Test: 10% fluorescein — The nasopharyngeal lesions were first identified endoscopically by nasal endoscope. Then, an initial dose of 0.5 mL prior to the examination with a maximum dose of 2.5 mL of 10% fluorescein (IV; Akorn Inc, Lake Forest, Illinois, USA) during the measurement procedure was defined according to the experiences of workgroup in the gastrointestinal tract.

SUMMARY:
To evaluate the use of probe-based confocal laser endomicroscopy (pCLE) in human nasopharyngeal mucosa for the differentiation of the nasopharyngeal squamous cell carcinomas.

DETAILED DESCRIPTION:
The aim of this study was to depict the applicability of pCLE examinations for diagnosing NPC in comparison to the gold standard of histopathological examination, as well as developed an easy-to-use and straightforward scoring system for the identification of NPC on the basis of morphological and architectural criteria in order to enable a valid and reproducible CLE assessment even for non-experts in their daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age
2. Indicated for nasal endoscope for indeterminate NPC
3. Willing and able to comply with study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

1. Subjects for whom pCLE procedures are contraindicated
2. Known allergy to fluorescein dye
3. If female, pregnant based on a positive hCG serum or an in vitro diagnostic test result or breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
pCLE classification and scoring system | 3 months
  Evaluation of pCLE diagnostic performance for the diagnosis of NPC when associated with other diagnostic information.

SECONDARY OUTCOMES:
the quantitative image analysis | 3 months
  Quantitative image features are calculated in the pCLE images

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, Phd &MD, Study Chair — Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No